CLINICAL TRIAL: NCT02998827
Title: Thalidomide Results in Diminished Ovarian Reserve in Reproductive Age Female IBD Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, pengxiang, Principal Investigator, Sixth Affiliated Hospital, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: E2016023
Record Dates: First submitted 2016-11-24; First posted 2016-12-20 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-12

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — Thalidomide; Infliximab; Azathioprine; Enteral Nutrition

ARMS (2):
- thalidomide (Experimental): use thalidomide tablet by mouth, every night for at least 6 months
  Interventions: Drug: Thalidomide
- other treatment (Active Comparator): the treatment include infliximab, azathioprine or enteral nutrition at least 6 months
  Interventions: Drug: infliximab, azathioprine; Other: enteral nutrition

INTERVENTIONS:
Drug: Thalidomide
  Arms: thalidomide
Drug: infliximab, azathioprine — other treatment include infliximab, azathioprine
  Arms: other treatment
Other: enteral nutrition
  Arms: other treatment

SUMMARY:
The effectiveness of thalidomide in treating inflammatory bowel disease has been widely recognized. Meanwhile, many serious adverse drug reactions were notified， but no reports on ovarian reserve function.Therefore, this study was to investigate the influence of thalidomide on function of ovarian reserve.

DETAILED DESCRIPTION:
It will be divided two groups of patients according to the treatment itself . One group was treated by thalidomide, the other was other treatment excluding. It will detect the function of ovarian reserve before and after treatment in both two groups, to investigate the influence of thalidomide on function of ovarian reserve.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50 years old Diagnosis of patients with CD

Exclusion Criteria:

* Pregnancy or lactation Period of women have fertility program during the study Treatment not foot eight weeks after last IFX Central or peripheral nerve disease Abnormal in liver and renal function Heart function failure Malignant tumor Active tuberculosis

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
difference AMH between thalidomide group and other treatment group | 1 year
  Anti-mullerian hormone（AMH）, as an important index to monitor the function of ovarian reserve, is majorly secreted by preantral follicles and antral follicles without fluctuation during menstrual cycle, not affected by hormone, and its change is earlier than sex hormone.
difference AFC between thalidomide group and other treatment group | 1 year
  The foundational follicles at 5- 10 mm of both ovaries were determined and the sum of antral follicles of both sides of ovaries was as antral follicles communicate (AFC)
difference E2 between thalidomide group and other treatment group | 1 year
  estradiol，a kind of hormone
difference FSH between thalidomide group and other treatment group | 1 year
  Follicle stimulating hormone,a kind of hormone